CLINICAL TRIAL: NCT00848471
Title: Validation of the Quark RMR Calorimeter (Cosmed) Versus Deltatrac II (GE Health Care Clinical Systems) for Measuring Energy Expenditure at Rest and in Dynamic Phase After a Meal in Adult Healthy and Obese Volunteers
Brief Title: Validation of the Quark RMR Calorimeter (Cosmed) Versus Deltatrac II (GE Health Care Clinical Systems)
Acronym: Protocol Quark
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Centre de Recherche en Nutrition Humaine Rhone-Alpe (Other)
Responsible Party: Pr Martine LAVILLE, Hôpital Edouard Herriot
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2008.539
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Healthy; Obesity
Keywords: Indirect calorimeter; Validation; Energy expenditure; Healthy volunteers
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Quark RMR calorimeter (Cosmed)
  Interventions: Device: Quark RMR
- 2 (Active Comparator): Deltatrac II (GE health Care Clinical Systems)
  Interventions: Device: Deltatrac II

INTERVENTIONS:
Device: Quark RMR — Quark RMR calorimeter (Cosmed)
  Arms: 1
Device: Deltatrac II — Deltatrac II (GE health Care Clinical Systems)
  Arms: 2

SUMMARY:
Measurement of energy expenditure at rest (12 hours fasting) and in dynamic phase after a meal (600kcal) to compare the results of the two calorimeters in standardized conditions for the validation of quark RMR versus Deltatrac II

DETAILED DESCRIPTION:
Clinically, energy expenditure is usually estimated using predictive equations, such as the Harris-Benedict equation, which consider the patient's weight, height, age and sex to determine energy needs. However these have been shown to be unsystematically incorrect and may vary by 70-140% when compared with indirect and direct calorimetry measurements.

That is why the most popular method of measurement of energy expenditure in research is via indirect calorimetry using a metabolic cart. Indirect calorimetry is the measurement of the volume of oxygen consumption and carbon dioxide production.

Actually, there are few numbers of indirect calorimeters available commercialy. The Deltatrac II metabolic cart was the gold standard. It has been extensively used in clinical research both for resting metabolic rate and substrate oxidation measurement during postprandial or an insulin clamp. The Quark RMR is also a metabolic cart too which was launched on the market to compete with the others calorimeters measuring resting metabolic rate.

As the Quark RMR and Deltatrac II use the same measure device (paramagnetic analyser for oxygen detection, infrared absorption for carbon dioxide detection) with the same sensitivity and time response according to constructor's data, we want to compare these two calorimeters for the measurement of energy expenditure and substrate oxidation at rest and during a meal in standardized conditions.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years old
* BMI between 20 and 35 kg/m²
* Weight stable for at least 2 months
* Safety subject during medical consultation
* Normal TSH -CRP -glycemia - creatinin

Exclusion Criteria:

* Medical or surgical history which may affect energy expenditure (renal -cardiovascular -hepatic- endocrine-inflamatory diseases)
* Drug use that could affect energy expenditure (steroids, nicotine substitutes, thyroid hormones)
* Eating disorder
* Intensive sportive activity (Baecke's score >5)
* Subjects who Smoke
* Claustrophobic subjects
* Pregnant women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
To compare the results obtained for the Deltatrac II and the Quark RMR for the measure of energy expenditure at rest in standardized conditions | At the end of the study

SECONDARY OUTCOMES:
To compare the results obtained for the Deltatrac II and the Quark RMR for the measure of energy expenditure after a food intake of 600kcal | At the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Martine LAVILLE, M.D, Principal Investigator — Hôpital Edouard Herriot
Locations (1):
- Centre de Recherche en Nutrition Rhône Alpes, Hôpital Edouard Herriot, Lyon, Rhone-Alps, France